CLINICAL TRIAL: NCT04642131
Title: The Effect of Fatigue, Caffeine Supplementation and Personalized Insoles on Biomechanics and Athletic Performance in Female Adult Soccer Players.
Brief Title: Effect of Caffeine Supplementation and Personalized Insoles on Females
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Were unable to recruit enough participants and the agreement with the laboratory providing the measurements stoped.
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Alejandro Gómez Bruton, Principal investigator, Universidad de Zaragoza
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: UZCUD2020-BIO-02
Record Dates: First submitted 2020-11-06; First posted 2020-11-24 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Caffeine; Fatigue; Injuries; Females Xy; Soccer; Biomechanical Parameters
Keywords: women; insoles; kinematics; kinetics; performance; athletics; team sport
MeSH Terms: conditions — Fatigue; Wounds and Injuries; Disorder of Sex Development, 46,XY

STUDY DESIGN:
Intervention Model Description: Participants will be given a bottle with either caffeine and carbohydrates or just carbohydrates, and personalized insoles or standard insoles. All participants will complete athletic and biomechanics tests before and after completing a 43 minute fatigue protocol.
Who Masked: Participant, Investigator
Masking Description: Participants will be given a bottle with either caffeine and carbohydrates or just carbohydrates.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Personalized insoles (Experimental): Personalized insoles without supplementation
  Interventions: Device: Personalized insoles
- Caffeine supplementation (Experimental): Standard insoles with caffeine supplementation (3mg/kg)
  Interventions: Dietary Supplement: Caffeine supplementation
- Control condition (Placebo Comparator): Standard insoles without supplementation
  Interventions: Other: Control condition

INTERVENTIONS:
Dietary Supplement: Caffeine supplementation — Participants will wear standard insoles and ingest caffeine in liquid form (3mg/kg) with carbohydrates.
  Arms: Caffeine supplementation
Device: Personalized insoles — Participants will wear personalized insoles and ingest a drink of carbohydrates without caffeine
  Arms: Personalized insoles
Other: Control condition — Participants will wear standard insoles and ingest a drink of carbohydrates without caffeine
  Arms: Control condition

SUMMARY:
Several studies have shown the positive effect that caffeine has on athletic performance related variables. Nonetheless, most studies have been developed in males and have not studied the possible effects on biomechanics and related injuries. Moreover, the inclusion of personalized insoles could also affect biomechanical patterns and thus injury incidence that has shown to be higher when athletes are fatigued. Therefore, the aim of the present randomized controlled trial is to evaluate the effect of fatigue, caffeine supplementation and personalized insoles on biomechanics and athletic performance in female adult soccer players.

ELIGIBILITY:
Inclusion Criteria:

* Females
* Soccer players who have been competing for at least 3 years

Exclusion Criteria:

* Participants with major injuries in the lower limbs within the 12 months before testing.
* Participants consuming ephedrine or related medicines

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2020-12-09 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Agility after fatigue and caffeine supplementation | One day
  Assessment of agility in seconds before and after a fatigue protocol is applied. Data will be collected with photoelectric cells.
Jump height after fatigue and caffeine supplementation | One day
  Assessment of jump height in centimetres before and after a fatigue protocol is applied. Data will be collected with force plates.
Repeated sprint ability after fatigue and caffeine supplementation | One day
  Assessment of repeated sprints ability in seconds before and after a fatigue protocol is applied. Data will be collected with photoelectric cells.
Agility after fatigue and personalized insoles | One day
  Assessment of agility in seconds before and after a fatigue protocol is applied. Data will be collected with photoelectric cells.
Jump height after fatigue and personalized insoles | One day
  Assessment of jump height in centimetres before and after a fatigue protocol is applied. Data will be collected with force plates.
Repeated sprint ability after fatigue and personalized insoles | One day
  Assessment of repeated sprints ability in seconds before and after a fatigue protocol is applied. Data will be collected with photoelectric cells.
Agility after fatigue and placebo | One day
  Assessment of agility in seconds before and after a fatigue protocol is applied. Data will be collected with photoelectric cells.
Jump height after fatigue and placebo | One day
  Assessment of jump height in centimetres before and after a fatigue protocol is applied. Data will be collected with force plates.
Repeated sprint ability after fatigue and placebo | One day
  Assessment of repeated sprints ability in seconds before and after a fatigue protocol is applied. Data will be collected with photoelectric cells.
Hip range of motion after fatigue and caffeine supplementation | During the intervention
  Assessment of hip range of motion in degrees assessed with VICON before and after a fatigue protocol is applied. Data will be collected with the VICON motion capture system.
Knee range of motion after fatigue and caffeine supplementation | During the intervention
  Assessment of knee range of motion in degrees assessed with VICON before and after a fatigue protocol is applied. Data will be collected with the VICON motion capture system.
Ankle range of motion after fatigue and caffeine supplementation | During the intervention
  Assessment of ankle range of motion in degrees assessed with VICON before and after a fatigue protocol is applied. Data will be collected with the VICON motion capture system.
Hip flexion moment after fatigue and caffeine supplementation | During the intervention
  Assessment of hip flexion moment in Nm·kg assessed with VICON before and after a fatigue protocol is applied. Data will be collected with the VICON motion capture system.
Knee flexion moment after fatigue and caffeine supplementation | During the intervention
  Assessment of knee flexion moment in Nm·kg assessed with VICON before and after a fatigue protocol is applied. Data will be collected with the VICON motion capture system.
Ankle flexion moment after fatigue and caffeine supplementation | During the intervention
  Assessment of ankle flexion moment in Nm·kg assessed with VICON before and after a fatigue protocol is applied. Data will be collected with the VICON motion capture system.
Hip range of motion after fatigue and personalized insoles | During the intervention
  Assessment of hip range of motion in degrees assessed with VICON before and after a fatigue protocol is applied. Data will be collected with the VICON motion capture system.
Knee range of motion after fatigue and personalized insoles | During the intervention
  Assessment of knee range of motion in degrees assessed with VICON before and after a fatigue protocol is applied. Data will be collected with the VICON motion capture system.
Ankle range of motion after fatigue and personalized insoles | During the intervention
  Assessment of ankle range of motion in degrees assessed with VICON before and after a fatigue protocol is applied. Data will be collected with the VICON motion capture system.
Hip flexion moment after fatigue and personalized insoles | During the intervention
  Assessment of hip flexion moment in Nm·kg assessed with VICON before and after a fatigue protocol is applied. Data will be collected with the VICON motion capture system.
Knee flexion moment after fatigue and personalized insoles | During the intervention
  Assessment of knee flexion moment in Nm·kg assessed with VICON before and after a fatigue protocol is applied. Data will be collected with the VICON motion capture system.
Ankle flexion moment after fatigue and personalized insoles | During the intervention
  Assessment of ankle flexion moment in Nm·kg assessed with VICON before and after a fatigue protocol is applied. Data will be collected with the VICON motion capture system.
Hip range of motion after fatigue and placebo | During the intervention
  Assessment of hip range of motion in degrees assessed with VICON before and after a fatigue protocol is applied. Data will be collected with the VICON motion capture system.
Knee range of motion after fatigue and placebo | During the intervention
  Assessment of knee range of motion in degrees assessed with VICON before and after a fatigue protocol is applied. Data will be collected with the VICON motion capture system.
Ankle range of motion after fatigue and placebo | During the intervention
  Assessment of ankle range of motion in degrees assessed with VICON before and after a fatigue protocol is applied. Data will be collected with the VICON motion capture system.
Hip flexion moment after fatigue and placebo | During the intervention
  Assessment of hip flexion moment in Nm·kg assessed with VICON before and after a fatigue protocol is applied. Data will be collected with the VICON motion capture system.
Knee flexion moment after fatigue and placebo | During the intervention
  Assessment of knee flexion moment in Nm·kg assessed with VICON before and after a fatigue protocol is applied. Data will be collected with the VICON motion capture system.
Ankle flexion moment after fatigue and placebo | During the intervention
  Assessment of ankle flexion moment in Nm·kg assessed with VICON before and after a fatigue protocol is applied. Data will be collected with the VICON motion capture system.

SECONDARY OUTCOMES:
Injury incidence | Six months
  Association between the primary outcomes and injury incidence registered through the International Federation of Association Football questionnaire (F-MARC)
Sleep disturbances after caffeine ingestion | Immediately after the intervention
  Rate of patients with sleep problems assessed with the Athens sleep questionnaire
Sleep disturbances after personalized insoles | Immediately after the intervention
  Rate of patients with sleep problems assessed with the Athens sleep questionnaire
Sleep disturbances after placebo | Immediately after the intervention
  Rate of patients with sleep problems assessed with the Athens sleep questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Zaragoza, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: Undecided